CLINICAL TRIAL: NCT01435148
Title: A Double Blind Randomised Pilot Study of Deep Brain Stimulation in Patients With Treatment Resistant Unipolar Major Depressive Disorder.
Brief Title: Deep Brain Stimulation in Treatment Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: North Bristol NHS Trust (Other)
Collaborators: University of Bristol (Other)
Responsible Party: Principal Investigator, Dr Andrea Malizia, Dr Andrea Malizia, North Bristol NHS Trust
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 1759; 06/Q2001/189 (Other: Bath NHS Research Ethics Committee)
Record Dates: First submitted 2011-09-02; First posted 2011-09-15 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Treatment Resistant Depression
Keywords: Deep Brain Stimulation; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Deep Brain Stimulation; Drug Implants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stimulation of SGC then VACNAC targets (Experimental): Stimulation of the subgenual cingulate cortex (SGC) target will take place first, followed by stimulation of the ventral anterior capsule nucleus accumbens target (VACNAC) if no clinical response after a minimum of 4 months.
  Interventions: Procedure: Deep Brain Stimulation, implanted
- Stimulation of VACNAC then SGC targets. (Experimental): Stimulation of the ventral anterior capsule nucleus accumbens target (VACNAC) will take place first, followed by stimulation of the subgenual cingulate cortex target (SGC) if no clinical response after a minimum of 4 months.
  Interventions: Procedure: Deep Brain Stimulation, implanted

INTERVENTIONS:
Procedure: Deep Brain Stimulation, implanted — Deep brain stimulator implanted during neurosurgery. Specific stimulation parameters programmed after surgery as required. After blinded study arms open stimulation of either or both targets.

SUMMARY:
Recurrent major depressive disorder affects about 3-5% of the population. It is anticipated that by 2020, depression will be the most common cause of disability worldwide in the 18-55 age group. About two-thirds of these patients respond to first-line treatment (antidepressants). In addition, prolonged administration of antidepressants in patients who respond results in remission in 80% of patients per year. However, a significant proportion of patients either fail to respond in spite of determined pharmacological treatments, electroconvulsive therapy and other treatments or do not achieve sustained remission. The personal, psychiatric, medical, social and economic consequences are devastating for these, treatment resistant, patients. This investigation aims to evaluate the feasibility of deep brain stimulation in patients with treatment resistant depression as a viable alternative to ablative neurosurgery.The hypothesis is that some patients will respond to stimulation in one site rather than the other and that some patients will respond to double rather than single site stimulation.

DETAILED DESCRIPTION:
Patients will be selected according to inclusion/ exclusion criteria after referral from their psychiatric team or, in exceptional cases, from their GP. Patients will be referred to the trial after being assessed by Dr Malizia (Consultant Senior Lecturer) in the Treatment Resistant Disorders Psychopharmacology clinic in the Bristol Royal Infirmary. Informed written consent and baseline measures will be taken for all patients.

We plan to recruit 8 patients with treatment resistant unipolar depression for a single blind trial of bilateral consecutive deep brain stimulation of Cg25 and ventral anterior capsule separately and then together. Medication will be left unchanged and maintained to the same level until the end of the study postoperatively. However, medication thought to be potentially detrimental in the long term will be stopped or reduced prior to surgery and a period of at least 6 weeks stability in prescribed medication will be required prior to baseline assessment.

The surgical procedure will be under general anaesthesia and will consist of implanting bilateral deep brain stimulating electrodes (four overall) into Brodmann's area 25 and the nucleus accumbens/ ventral anterior capsule. Following the operation a period of one-week recovery will be allowed to minimise any effect secondary to target impact effect at surgery or from post-operative oedema.

After recovery the combination of electrodes with maximal response will be assessed in a double blind design (patient and raters).

Stimulation will be bilateral. Four patients will be randomised to receive Cg25 stimulation first and 4 patients will be randomised to receive anterior capsule/ventral striatal stimulation first. Patients will be blind to the order of stimulation, to the contacts selected and to any 'off' period in the contact selection process.

After at least four months patients will crossover to the alternative site of stimulation unless they have achieved remission (MADRS <8 for at least two months). Patients and raters will still be blind to the site of stimulation. After a further four months selection will be for both sets of contacts that have achieved best results. If the MADRS score is <8 with one location and no significant improvement has occurred in the other (MADRS>18 and improvement <25%), then only one set of contacts will be stimulated from there on.

Clinical assessments will be at least two monthly on average.

The full evaluation procedure will last an average of 18 months from surgical implantation of the electrodes.

ELIGIBILITY:
Inclusion Criteria:

Patients who have major depressive disorder (according to the Diagnostic and Statistical Manual version IV) and who:

1. Do not respond or have ceased to respond to treatment including:

   * Cognitive Behaviour Therapy (CBT) or other validated psychotherapy.
   * Antidepressants from three different classes in BNF or maximum tolerated (if lower than BNF) doses
   * Lithium augmentation
   * 2 courses of ECT (or only respond to "maintenance" ECT)(lack of response in previous episodes and unwillingness to try again will also count).
2. Consent to take part in the trial
3. Are physically fit
4. Have no suicidal intent
5. Have no history of hypomania, mania or psychosis
6. Montgomery Asberg Depression Rating Scale score > 21

Exclusion Criteria:

1. Patients with a history of continuous depression from late teens or early twenties without clear response to treatments or without periods of spontaneous remission,
2. Pregnancy
3. History of significant head trauma
4. Dementia
5. Cerebral infarcts
6. Poor physical health
7. No capacity to consent
8. Inability to carry out research protocol
9. Mood incongruent psychotic phenomena or drug or alcohol addiction. In addition patients will be excluded if detained under the Mental Health Act.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Decrease in Montgomery and Asberg Rating Scale score of at least 50% at an average of 18 months after implantation. | End of contact selection and adjustment plus 6 months. An average of 18 months after implantation.
  MADRS is a standard depression rating scale for major depressive disorder over time

SECONDARY OUTCOMES:
Clinical Global Impression Improvement Scale(CGI-I). Score <4. | End of contact selection and adjustment plus 6 months. An average of 18 months after implantation
  The Clinical Global Impression Scale (CGI) will be used to asses global functioning over time in our patients and will be completed by the interviewing psychiatrist.
Global Assessment of Functioning scale, an improvement of >1/2(100-initial score) | End of contact selection and adjustment plus 6 months. An average of 18 months after implantation
  The Global Assessment of Functioning scale is a standardized scale used to asses functioning in patients with chronic conditions. It is useful here as it allows an aspect of 'social' functioning to be assessed during the study. It will be completed by the interviewing psychiatrist.
A decrease of 50% in Hamilton Depression Rating Scale (17 items) at End of contact selection and adjustment plus 6 months. An average of 18 months after implantation | End of contact selection and adjustment plus 6 months. An average of 18 months after implantation
  Ham_D is a standard observer rated measure of depression in major depressive disorder over time

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Malizia, MD, PhD, Principal Investigator — Bristol University
Locations (1):
- Neurosurgey Department, Frenchay Hospital, Bristol, Bristol, United Kingdom